CLINICAL TRIAL: NCT07052188
Title: Evaluation of the Effect of Preoperative Stenting Duration on Stone-Free Rates and the Need for Secondary Surgical Intervention in Retrograde Intrarenal Surgery
Brief Title: Effect of Preop Stent Duration on SFR and Secondary Intervention in RIRS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bedreddin Kalyenci (Other)
Responsible Party: Sponsor-Investigator, Bedreddin Kalyenci, Principal Investigator, Adiyaman University
Organization: Adiyaman University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRÜ/24.21.46
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Stone, Urinary; Stone, Kidney
Keywords: Ureteral stent; retrograde intrarenal surgery; prestenting; preoperative ureteral stenting
MeSH Terms: conditions — Urinary Calculi; Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients will have RIRS without any preoperative double J (DJ) stenting (Experimental)
  Interventions: Procedure: without any preoperative stenting
- Patients will have a double-J (DJ) stent placed with sedation and undergo RIRS within 2-4 weeks. (Experimental)
  Interventions: Procedure: (DJ) stent placed with sedation and undergo RIRS within 2-4 weeks
- Patients will have a DJ stent placed with sedation and undergo RIRS within 4-6 weeks. (Experimental)
  Interventions: Procedure: Patients will have a DJ stent placed with sedation and undergo RIRS within 4-6 weeks.

INTERVENTIONS:
Procedure: without any preoperative stenting — Patients will have RIRS without any preoperative stenting.
  Arms: Patients will have RIRS without any preoperative double J (DJ) stenting
Procedure: (DJ) stent placed with sedation and undergo RIRS within 2-4 weeks — Patients will have a double-J (DJ) stent placed with sedation and undergo RIRS within 2-4 weeks.
  Arms: Patients will have a double-J (DJ) stent placed with sedation and undergo RIRS within 2-4 weeks.
Procedure: Patients will have a DJ stent placed with sedation and undergo RIRS within 4-6 weeks. — Patients will have a DJ stent placed with sedation and undergo RIRS within 4-6 weeks
  Arms: Patients will have a DJ stent placed with sedation and undergo RIRS within 4-6 weeks.

SUMMARY:
This study aims to evaluate how placing a stent before surgery (preoperative stenting or passive dilation) affects the success rate of retrograde intrarenal surgery (RIRS), which is performed for kidney stones. Specifically, we will examine whether stenting improves the chance of becoming stone-free after surgery and reduces the need for a second surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with an indication for RIRS (Retrograde Intrarenal Surgery)

Exclusion Criteria:

* Patients under 18 or over 65 years of age
* Patients who cannot be followed up in the postoperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with stone-free | in the first month after surgery
Number of Participants with additional surgery was needed | in the first month after surgery

SECONDARY OUTCOMES:
Number of Participants with postoperative complications | within 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Adıyaman University, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after the completion of the study